CLINICAL TRIAL: NCT00736086
Title: A Post-Market, Prospective, Multi-Center, Study to Evaluate Safety and Efficacy of the StarClose™ Vascular Closure System in Patients Who Are Ambulated Early Post-Diagnostic Catheterization
Brief Title: RISE: A Clinical Evaluation of the StarClose™ Vascular Closure System
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Boris Jelecic, Abbott Vascular
Other Study IDs: AVD-640-0057
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Last update posted 2008-08-15 (Estimated); Status verified 2008-08

CONDITIONS: Peripheral Vascular Disease; Cardiovascular Disease
Keywords: femoral artery; post-percutaneous cardiac catheterization; post-percutaneous peripheral vascular catheterization; post-percutaneous diagnostic catheterization; early ambulation; vascular closure
MeSH Terms: conditions — Peripheral Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Subjects who are ambulated early post-percutaneous, cardiac or peripheral vascular, diagnostic catheterization procedures with the use of StarClose® Vascular Closure System in the femoral artery after diagnostic catheterization procedure.
  Interventions: Device: Vessel Closure (StarClose™)

INTERVENTIONS:
Device: Vessel Closure (StarClose™)

SUMMARY:
To evaluate early ambulation in patients who receive the StarClose™ VCS post-percutaneous diagnostic procedure.

DETAILED DESCRIPTION:
To evaluate the StarClose™ VCS in the femoral artery in subjects who are ambulated early post-percutaneous cardiac or peripheral vascular, diagnostic catheterization procedure. The clinical use of vascular closure devices for rapid hemostasis after femoral access was first reported in 1991. 18 participants may be ambulated almost immediately after diagnostic coronary angiography and discharged many hours earlier than currently practiced in most centers utilizing a supine restriction period of 6 hours after diagnostic catheterization.14 After coronary interventions, participant comfort is additionally increased by immediate sheath removal.

This early ambulation study is an evaluation of a clip-based technology, which achieves vascular hemostasis with the use of a novel extravascular Nitinol clip to provide an immediate mechanical closure that does not depend upon the body's clotting system. The procedures will be performed in participants who meet specific entrance criteria.

ELIGIBILITY:
Inclusion:

* Subject must be 18-85.
* Subject must be an acceptable candidate for an elective,non-emergent diagnostic procedure performed percutaneously via the common femoral artery through either a 5F or 6F procedural sheath.
* Subject is an acceptable candidate for emergent vascular surgery.
* Subject agrees to follow-up evaluations to assess for complications related to femoral access site.
* If among the 50 ultrasound sub-study Subjects enrolled,Subject agrees to have an ultrasound of femoral artery performed post-procedure during the 30 ± 7 days follow-up visit.
* Subject or legal representative has been informed of the nature of the study and agrees to provisions and has provided written informed consent as approved by the Institutional Review Board of respective clinical site.

Exclusion:

* History of bleeding diathesis or coagulopathy including hemophilia, von Willebrand's disease, and/or a current, known platelet count <100,000 cells/mm3, or baseline INR > 1.7.
* Body Mass Index (BMI) ³ 35 kg/m2.
* Presence of significant anemia (Hgb < 10 g/dL, Hct < 30%).
* Advanced Subject refusal of blood transfusions, should transfusion become necessary.
* Participation in another trial of an investigational drug or device that has not yet completed follow-up requirements.
* Pregnant or lactating female.
* Clinically severe peripheral vascular disease in the ipsilateral limb, defined as severe claudication (walking < 100 feet), weak or absent pulses, or lower extremity vascular graft.
* History of ipsilateral femoral arterial puncture within previous three months or history of vascular closure device deployment in ipsilateral femoral artery at any time.
* Subject has unilateral or bilateral lower extremity amputation(s).
* Subject is unable to routinely walk at least 20 feet without assistance.
* Subject has an active systemic or cutaneous infection or inflammation.
* Subject has a pre-existing severe non-cardiac systemic disease or illness with a life expectancy of < 30 days.
* Subject has already participated in this Study.
* Subject has known allergy to nitinol.

Access Site Exclusion-(*Evaluated via Limited Femoral Angiogram)

* Pseudoaneurysm or AV fistula present in ipsilateral femoral artery prior to arterial closure.*
* Puncture distal to the common femoral artery bifurcation or above the inguinal ligament which is typically defined by the inferior border of the inferior epigastric artery on sheath angiogram or the upper third of the femoral head by plain fluoroscopy.*
* The arterial lumen diameter at the arteriotomy site is < 5mm by visual estimate.*
* Angiographic evidence of calcified lesions at the arteriotomy site.*
* Difficulty inserting the introducer sheath at the start of the catheterization procedure due to vessel scarring or tortuosity, or anterior/posterior wall femoral artery punctures or greater than 2 ipsilateral arterial puncture attempts at the time of the percutaneous procedure.
* Known iliac or femoral stenosis >50% or previous bypass surgery or stent placement in the vicinity of the puncture site.
* Planned percutaneous procedure (diagnostic or intervention) in ipsilateral femoral artery prior to the 30-day follow-up evaluation.
* Subject has intra-procedural bleeding around the access site.
* Presence or previous use of an intra-aortic balloon pump through the existing arterial puncture site.

Procedural Exclusion:

* Low molecular weight heparin administration within 8 hours of enrollment.
* For cases where anticoagulants are used, ACT level > 350 seconds at time of enrollment.
* Subject is determined to require treatment that will extend hospitalization (e.g. ---Subject is undergoing CABG surgery or staged PTCA).
* Persistent hypertension (SBP >180 or DBP >110 mm Hg) unresponsive to medical -therapy at time of enrollment.
* Placement of an ipsilateral femoral venous sheath during procedure.
* Presence of clinically significant hematoma (> 6 cm) in ipsilateral femoral artery prior to arterial closure.
* Placement of introducer sheath < 5F or > 6F during procedure.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are ambulated early post-percutaneous, cardiac or peripheral vascular, diagnostic catheterization procedure
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2006-03; Primary Completion 2006-11 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Kussmaul, MD, Principal Investigator — Drexel University/Hahnemann
Locations (11):
- United States (11):
  - Scripps Memorial Hospital, La Jolla, California
  - Fuqua Heart Center/ Piedmont Hospital, Atlanta, Georgia
  - Heart Care Midwest (OSF/St Francis), Peoria, Illinois
  - The Care Group LLC (St. Vincent's Hospital), Indianapolis, Indiana
  - Bay Regional Medical Center, Bay City, Michigan
  - Minneapolis Heart Institute Foundation/Abbott Northwestern Hospital, Minneapolis, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - New York Methodist Hospital, Brooklyn, New York
  - Buffalo Heart group, Buffalo, New York
  - North Ohio Research LTD Elyria Regional Medical, Elyria, Ohio
  - Drexel University College of Medicine Hahnemann, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Krone RJ, Johnson L, Noto T. Five year trends in cardiac catheterization: a report from the Registry of the Society for Cardiac Angiography and Interventions. Cathet Cardiovasc Diagn. 1996 Sep;39(1):31-5. doi: 10.1002/ccd.1810390102. PMID 8874942
- [Background] Waksman R, Scott NA, Ghazzal ZM, Mays R, Frerichs FA, Petersen JY, King SB 3rd. Randomized comparison of flexible versus nonflexible femoral sheaths on patient comfort after angioplasty. Am Heart J. 1996 Jun;131(6):1076-8. doi: 10.1016/s0002-8703(96)90079-4. PMID 8644584
- [Background] Bogart DB, Bogart MA, Miller JT, Farrar MW, Barr WK, Montgomery MA. Femoral artery catheterization complications: a study of 503 consecutive patients. Cathet Cardiovasc Diagn. 1995 Jan;34(1):8-13. doi: 10.1002/ccd.1810340304. PMID 7728861
- [Background] Christensen B, Lacarella C, Manion R, Bruhn-Ding B, Meyer S, Wilson R. Sandbags do not prevent complications after catheterization. Circulation 90:I-205, 1994.
- [Background] Pracyk JB, Wall TC, Longabaugh JP, Tice FD, Hochrein J, Green C, Cox G, Lee K, Stack RS, Tcheng JE. A randomized trial of vascular hemostasis techniques to reduce femoral vascular complications after coronary intervention. Am J Cardiol. 1998 Apr 15;81(8):970-6. doi: 10.1016/s0002-9149(98)00074-5. PMID 9576155
- [Background] Resar JR, Prewitt KC, Wolff MR, Blumenthal R, Raqueno JV, Brinker JA. Percutaneous transluminal coronary angioplasty through 6F diagnostic catheters: a feasibility study. Am Heart J. 1993 Jun;125(6):1591-6. doi: 10.1016/0002-8703(93)90745-u. PMID 8498298
- [Background] Cragg AH, Nakagawa N, Smith TP, Berbaum KS. Hematoma formation after diagnostic angiography: effect of catheter size. J Vasc Interv Radiol. 1991 May;2(2):231-3. doi: 10.1016/s1051-0443(91)72287-2. PMID 1799761
- [Background] Waksman R, King SB 3rd, Douglas JS, Shen Y, Ewing H, Mueller L, Ghazzal ZM, Weintraub WS. Predictors of groin complications after balloon and new-device coronary intervention. Am J Cardiol. 1995 May 1;75(14):886-9. doi: 10.1016/s0002-9149(99)80681-x. PMID 7732995
- [Background] Campeau L. Percutaneous radial artery approach for coronary angiography. Cathet Cardiovasc Diagn. 1989 Jan;16(1):3-7. doi: 10.1002/ccd.1810160103. PMID 2912567
- [Background] Kiemeneij F, Laarman GJ, Odekerken D, Slagboom T, van der Wieken R. A randomized comparison of percutaneous transluminal coronary angioplasty by the radial, brachial and femoral approaches: the access study. J Am Coll Cardiol. 1997 May;29(6):1269-75. doi: 10.1016/s0735-1097(97)00064-8. PMID 9137223
- [Background] Bertrand ME, Legrand V, Boland J, Fleck E, Bonnier J, Emmanuelson H, Vrolix M, Missault L, Chierchia S, Casaccia M, Niccoli L, Oto A, White C, Webb-Peploe M, Van Belle E, McFadden EP. Randomized multicenter comparison of conventional anticoagulation versus antiplatelet therapy in unplanned and elective coronary stenting. The full anticoagulation versus aspirin and ticlopidine (fantastic) study. Circulation. 1998 Oct 20;98(16):1597-603. doi: 10.1161/01.cir.98.16.1597. PMID 9778323
- [Background] Leon MB, Baim DS, Popma JJ, Gordon PC, Cutlip DE, Ho KK, Giambartolomei A, Diver DJ, Lasorda DM, Williams DO, Pocock SJ, Kuntz RE. A clinical trial comparing three antithrombotic-drug regimens after coronary-artery stenting. Stent Anticoagulation Restenosis Study Investigators. N Engl J Med. 1998 Dec 3;339(23):1665-71. doi: 10.1056/NEJM199812033392303. PMID 9834303
- [Background] Dick RJ, Popma JJ, Muller DW, Burek KA, Topol EJ. In-hospital costs associated with new percutaneous coronary devices. Am J Cardiol. 1991 Oct 1;68(9):879-85. doi: 10.1016/0002-9149(91)90403-8. PMID 1927947
- [Background] Krause PB, Klein LW. Utility of a percutaneous collagen hemostasis device: to plug or not to plug? J Am Coll Cardiol. 1993 Nov 1;22(5):1280-2. doi: 10.1016/0735-1097(93)90530-e. No abstract available. PMID 8227780
- [Background] Anderson HV, Bertrand M, Whitworth HB, Sax FL, Willerson JT for the Restore Investigators. Bleeding risk with platelet inhibition using Tirofiban: The Restore Trial. Circulation. 94:I-553, 1996.
- [Background] Lincoff AM, Tcheng JE, Miller DP, Booth JE, Montague EA, Topol EJ. Marked enhancement of clinical efficacy of platelet GP IIb/IIIa blockade with c7E3Fab (Abciximab) linked to reduction in bleeding complications: Outcome in the EPILOG and EPIC trials. Circulation 94:I-375, 1996.
- [Background] Goods CM, Liu MW, Jain SP, Mathur A, Yadav JS, Al-Shalbi KF, Dean LS, Iyer SS, Parks JM, Roubin GS. Low molecular weight heparin versus standard heparin in participants at high risk for stent thrombosis: Clinical outcomes. Circulation 94:I-684, 1996.
- [Background] Ernst S, Kloss R, Schräder R, Kaltenbach M, Sigwart U, Sanborn TA. Immediate sealing of arterial puncture sites after catheterization and PTCA using a vascular hemostasis device with collagen: an international study. Circulation 84:I-272, 1991.
- [Background] Silber S, Dorr R, Muhling H, Konig U. Sheath pulling immediately after PTCA: comparison of two different deployment techniques for the hemostatic puncture closure device: a prospective, randomized study. Cathet Cardiovasc Diagn. 1997 Aug;41(4):378-83. doi: 10.1002/(sici)1097-0304(199708)41:43.0.co;2-2. PMID 9258477
- [Background] Silber S. Rapid hemostasis of arterial puncture sites with collagen in patients undergoing diagnostic and interventional cardiac catheterization. Clin Cardiol. 1997 Dec;20(12):981-92. doi: 10.1002/clc.4960201203. PMID 9422835
- [Background] Silber S. Hemostasis success rates and local complications with collagen after femoral access for cardiac catheterization: analysis of 6007 published patients. Am Heart J. 1998 Jan;135(1):152-6. doi: 10.1016/s0002-8703(98)70356-4. PMID 9453535
- [Background] Hoffer EK, Bloch RD. Percutaneous arterial closure devices. J Vasc Interv Radiol. 2003 Jul;14(7):865-85. doi: 10.1097/01.rvi.0000071086.76348.8e. PMID 12847195
- [Background] Duffin DC, Muhlestein JB, Allisson SB, Horne BD, Fowles RE, Sorensen SG, Revenaugh JR, Bair TL, Lappe DL. Femoral arterial puncture management after percutaneous coronary procedures: a comparison of clinical outcomes and patient satisfaction between manual compression and two different vascular closure devices. J Invasive Cardiol. 2001 May;13(5):354-62. PMID 11385148
- [Background] Shammas NW, Rajendran VR, Alldredge SG, Witcik WJ, Robken JA, Lewis JR, McKinney D, Hansen CA, Kabel ME, Harris M, Jerin MJ, Bontu PR, Dippel EJ, Labroo A. Randomized comparison of Vasoseal and Angioseal closure devices in patients undergoing coronary angiography and angioplasty. Catheter Cardiovasc Interv. 2002 Apr;55(4):421-5. doi: 10.1002/ccd.10098. PMID 11948884
- [Background] Ward SR, Casale P, Raymond R, Kussmaul WG 3rd, Simpfendorfer C. Efficacy and safety of a hemostatic puncture closure device with early ambulation after coronary angiography. Angio-Seal Investigators. Am J Cardiol. 1998 Mar 1;81(5):569-72. doi: 10.1016/s0002-9149(97)00970-3. PMID 9514451
- [Background] Kussmaul WG 3rd, Buchbinder M, Whitlow PL, Aker UT, Heuser RR, King SB, Kent KM, Leon MB, Kolansky DM, Sandza JG Jr. Rapid arterial hemostasis and decreased access site complications after cardiac catheterization and angioplasty: results of a randomized trial of a novel hemostatic device. J Am Coll Cardiol. 1995 Jun;25(7):1685-92. doi: 10.1016/0735-1097(95)00101-9. PMID 7759724
- [Background] Kapadia SR, Raymond R, Knopf W, Jenkins S, Chapekis A, Ansel G, Rothbaum D, Kussmaul W, Teirstein P, Reisman M, Casale P, Oster L, Simpfendorfer C. The 6Fr Angio-Seal arterial closure device: results from a multimember prospective registry. Am J Cardiol. 2001 Mar 15;87(6):789-91, A8. doi: 10.1016/s0002-9149(00)01507-1. PMID 11249907
- [Derived] Burke MN, Hermiller J, Jaff MR. StarClose vascular closure system (VCS) is safe and effective in patients who ambulate early following successful femoral artery access closure--results from the RISE clinical trial. Catheter Cardiovasc Interv. 2012 Jul 1;80(1):45-52. doi: 10.1002/ccd.23176. Epub 2011 Dec 8. PMID 22162141